CLINICAL TRIAL: NCT01500499
Title: The Role of AF1q in Progression of Leukemia
Brief Title: Role of Biomarkers in Disease Progression in Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML12B2; COG-AAML12B2 (Other: Children's Oncology Group); AAML12B2 (Other: Children's Oncology Group); NCI-2012-00099 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-12-24; First posted 2011-12-28 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia; childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Gene Expression Profiling; Gene Rearrangement; Polymerase Chain Reaction; Blotting, Western; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: gene rearrangement analysis
Genetic: polymerase chain reaction
Genetic: protein analysis
Genetic: western blotting
Other: laboratory biomarker analysis
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of blood, tissue, and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies the role of biomarkers in disease progression in samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the subcellular localization of the MLL-AF1q fusion protein in leukemia cells.

OUTLINE: Cryopreserved specimens are analyzed for MLL-AF1q fusion protein and AF1 gene expression by mass spectrometry, western blot analysis, semi-quantitative PCR, and qPCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cryopreserved acute myeloid leukemia specimens

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Subcellular localization of the MLL-AF1q fusion protein in leukemia cells

CONTACTS AND LOCATIONS:
Overall Officials: Julie D. Saba, MD, PhD, Principal Investigator — UCSF Benioff Children's Hospital Oakland